CLINICAL TRIAL: NCT02176551
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Product 0405 To A Vehicle Control In The Treatment Of Mild To Moderate Atopic Dermatitis In Pediatric Subjects
Brief Title: Study Comparing Product 0405 to a Vehicle Control in the Treatment of Mild to Moderate Atopic Dermatitis in Pediatric Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0405-01-06
Record Dates: First submitted 2014-06-17; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Product 0405 (Experimental): Topical active investigational Product 0405
  Interventions: Drug: Product 0405
- Placebo for Product 0405 (Placebo Comparator): Topical Placebo for Product 0405
  Interventions: Drug: Placebo for Product 0405

INTERVENTIONS:
Drug: Product 0405 — Product 0405 will be administered topically twice daily for 28 days.
  Arms: Product 0405
Drug: Placebo for Product 0405 — Placebo for Product 0405 will be administered topically twice daily for 28 days.
  Arms: Placebo for Product 0405

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of product 0405 in pediatric subjects with Mild to Moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
Treatment medication will be administered topically twice daily for 28 days

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Atopic Dermatitis
* Good health with the exception of Atopic Dermatitis
* Percent body surface area minimum requirements

Exclusion Criteria:

* Subjects who are pregnant, nursing or planning a pregnancy

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Statistically significant superiority of the test Product 0405 to the vehicle | 28 days
  Statistically significant superiority of the test Product 0405 to the vehicle

SECONDARY OUTCOMES:
Incidence of success based on the Investigators Static Global Assessment and the Clinical Signs and Symptoms (erythema, scaling) at the end of treatment. | 28 days
  Incidence of success based on the Investigators Static Global Assessment and the Clinical Signs and Symptoms (erythema, scaling) at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Kaplan, Study Director — Fougera Pharmaceuticals Inc.